CLINICAL TRIAL: NCT00202787
Title: Open-label, Phase II, Randomised, Pilot Study to Evaluate the Safety and Efficacy of Combination Therapy With Cetuximab and FOLFOX4 or FOLFOX4 Alone in Patients Colorectal Cancer and Initially Non-resectable
Brief Title: Safety and Efficacy Study of Combination Therapy With Cetuximab and FOLFOX4 in Patients With Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTD-04-02; eudract-number: 2004-001700-12
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; cetuximab; FOLFOX4
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): FOLFOX-4+cetuximab
  Interventions: Drug: FOLFOX-4+cetuximab
- 2 (Active Comparator): FOLFOX-4
  Interventions: Drug: FOLFOX-4

INTERVENTIONS:
Drug: FOLFOX-4+cetuximab — Cetuximab; Weekly administration of Cetuximab IV (initial infusion of 400 mg/m2 for 120 minutes followed by subsequent maintenance doses of 250 mg/m2 for 60 minutes);
  FOLFOX-4: Every two week Oxaliplatin; 85 mg/m2 ; day 1 Folinic acid; 200 mg/m2 ; day 1 and 2 5-FU ; Bolus 400 mg/m2 + CI 600 mg/m2 22 h day 1 and 2
  Arms: 1
Drug: FOLFOX-4 — FOLFOX-4: Every two week Oxaliplatin; 85 mg/m2 ; day 1 Folinic acid; 200 mg/m2 ; day 1 and 2 5-FU ; Bolus 400 mg/m2 + CI 600 mg/m2 22 h day 1 and 2
  Arms: 2

SUMMARY:
The purpose of this study is to determine confirmed objective response rate to combination therapy with cetuximab and FOLFOX4 or FOLFOX4 alone in patients with CRC and non-resectable hepatic metastases

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Men and women < 75 years
* Histologically confirmed diagnosis of CRC
* Metastatic colorectal carcinoma with exclusive non-resectable hepatic metastases, due to fulfillment of one of the following criteria:

  1. Number of hepatic metastases > or= 4;
  2. Size of one or more hepatic metastases > 5 cm diameter;
  3. Vascular involvement and/or poor site that prevent complete resection of hepatic disease and/or require resection with the remaining liver mass less than 25-30% of functional liver.
* Presence of at least one lesion detectable by two-dimensional measurement.
* Karnofsky functional status >or=70% at the time of enrollment in study
* Life expectancy greater than 3 months.
* Patients must not have received chemotherapy for advanced/metastatic disease.
* Patients with the following characteristics will be enrolled:

  1. Recurrence after adjuvant treatment with 5-fluorouracil/folinic acid or capecitabine +/- radiotherapy with disease-free period > 6 months following conclusion of treatment.
  2. Recurrence after surgical and/or radiotherapy treatment without adjuvant systemic treatment.
  3. De novo diagnosis of disease.
* Proper liver function, defined by aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) < or = 2.5 x ULN (< or = 5 x ULN if there are hepatic metastases) and total bilirubin count < 1.5 x ULN.
* Proper kidney function, defined as serum creatinine < 1.5 x ULN.
* Proper hematological function, defined as neutrophil count > or = 1.5 x 109/l , platelets > or = 100 X 109/l and hemoglobin > or = 9 g/dl.
* Effective birth control method for men as well as women if there is possibility of pregnancy

Exclusion Criteria:

* Documented or suspected cerebral and/or leptomeningeal metastases.
* Metastasis in any other non-hepatic site, including extrahepatic lymph node metastases.
* Surgery (excluding biopsy for diagnosis) and/or radiotherapy within 4 weeks prior to enrollment in the study.
* Participation in another clinical trial with medication in the past 30 days.
* Chronic, concomitant administration of systemic immunotherapy, chemotherapy, hormone therapy or any other investigational drug.
* Prior malignant tumour in past 5 years, except history of basal cell skin carcinoma or pre-invasive cervical carcinoma.
* Any investigational drug during the 4 weeks prior to enrolment.
* Prior administration of monoclonal antibodies, EGFR signal transduction inhibitors or EGFR-targeted treatment.
* Prior participation in study in which treatment with cetuximab can be assigned (whether or not treatment with cetuximab is received)
* Acute or subacute intestinal occlusion or history of inflammatory intestinal disease.
* Evidence of grade 3 or 4 allergic reaction to any of the treatment components.
* Clinically relevant peripheral neuropathy.
* Clinically relevant myocardial disease or history of myocardial infarction in the past 12 months.
* Known abuse of alcohol / drugs, Legal incapacity or limited legal capacity.
* Any medical or psychological disorder which, in the opinion of the investigator, does not allow the patient to conclude the study or sign the informed consent.
* Pregnant or nursing woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2005-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Determine confirmed objective response rate | 2005-2009

SECONDARY OUTCOMES:
Determine safety of combination, surgical resectability and R0 resections, clinical benefit, time to disease progression, time to onset of response, duration of response, time to treatment failure, overall survival time | 2005-2009
determination of polymorphisms of the intron 1 of the EGFR gene, TS, XRCC1, XPD, serum levels of EGFR and ATP7A and ATP7B, nº of copies of EGFR gene, the levels of PTEN, EGFR, AKT y MAPK proteins, and mutations at EGFR, PI3KCA, K-RAS y B-RAF genes | 2005-2009

CONTACTS AND LOCATIONS:
Overall Officials: Albert Abad, Study Chair — Spanish Cooperative Group for Gastrointestinal Tumour Therapy (TTD)
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy (TTD), Madrid, Spain